CLINICAL TRIAL: NCT05065073
Title: Iso-Osmolar vs. Low-Osmolar Contrast Agents for Optical Coherence Tomography
Acronym: GE OCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE OCT
Record Dates: First submitted 2021-09-14; First posted 2021-10-01 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease; Contrast Media Reaction
Keywords: Optical Coherence Tomography; Contrast Agents
MeSH Terms: conditions — Coronary Artery Disease | interventions — iodixanol; Iohexol

STUDY DESIGN:
Intervention Model Description: Randomized, controlled study. Each patient will be randomized to undergoing OCT image acquisition with iso-osmolar contrast media first, or with low-osmolar contrast media first. Following this will be a second OCT image acquisition of the same coronary vessel with the other contrast media. Thus, each patient will serve as comparator to themselves, and to each other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iso-Osmolar Contrast Media (Active Comparator): Will receive iso-osmolar media first, low-osmolar media second
  Interventions: Drug: Iodixanol; Drug: Iohexol
- Low-Osmolar Contrast Media (Active Comparator): Will receive low-osmolar media first, iso-osmolar media second
  Interventions: Drug: Iodixanol; Drug: Iohexol

INTERVENTIONS:
Drug: Iodixanol — Iso-osmolar Contrast Media
  Other Names: Visipaque
Drug: Iohexol — Low-Osmolar Contrast Media
  Other Names: Omnipaque

SUMMARY:
The proposed study aims to compare (a) volume contrast administered for Optical Coherence Tomography (OCT) Imaging, (b) length of clear OCT images, and (c) electrocardiographic changes immediately after contrast injection between iso-osmolar and low-osmolar contrast agents. The proposed study is a prospective, single-centered, randomized controlled, study that will compare an iso-osmolar vs. a low-osmolar contrast agent in patients undergoing clinically indicated coronary OCT imaging. Each patient will be randomized to OCT acquisition.

DETAILED DESCRIPTION:
Patients referred to the Cardiac Catheterization laboratory for clinically indicated coronary angiography and coronary OCT imaging will be identified by a study team member and screened for eligibility. The proposed study is a prospective, single-center, randomized, controlled, study that will compare an iso-osmolar vs a low-osmolar contrast agent in patients undergoing clinically-indicated coronary OCT imaging. Each patient will be randomized to OCT acquisition. Eligible patients will be approached to obtain informed consent by a member of the study team. Once consent is obtained and inclusion and exclusion criteria are verified, patients are randomized to undergoing OCT image acquisition with iso-osmolar contrast media(IOCM) first or with low-osmolar contrast media first (LOCM).

Then the patients undergo coronary angiography and OCT imaging as per clinical standard of care. However, during the OCT imaging acquisition based on their randomization assignment the patient will undergo the 1st OCT imaging run with either iso-osmolar contrast media or with low-osmolar contrast media. Following this a 2nd OCT imaging run of the same coronary vessel will be done using the other contrast media that was not used during the first run. Therefore, each patient will serve as a comparator to themselves, but also to each other. The electrocardiogram will be recorded during and for 30 seconds after each injection and analyzed offline for detection of any changes

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or greater
2. Willing and able to give informed consent. The patients must be able to comply with study procedures
3. Undergoing clinically-indicated coronary angiography and OCT

Exclusion Criteria

1. Baseline electrocardiographic changes hindering interpretation (such as left bundle-branch block, and >1 mm ST segment depression)
2. Emergency cardiac catheterization (for example in patients with ST-segment elevation acute myocardial infarction)
3. Inability to provide symptomatic assessment
4. Known allergy to contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Contrast Volume after Injection | 30 seconds after injection
  Contrast volume will be measured after each injection

SECONDARY OUTCOMES:
Clear OCT Images | Intra-operative
  Length of clear OCT images will be defined as visible lumen border >270 degrees
Electrocardiographic (ECG) Changes | During and 30 seconds after injection
  Electrocardiographic(ECG) changes will be assessed during and for a period of 30 seconds after each injection of contrast for OCT, to detect and quantify any of the following abnormalities: arrhythmias, mean axis deviation and QRS enlargement (type A abnormalities); and ventricular repolarization (ST/T) changes (type B abnormalities)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil Brilakis, MD, PhD, Principal Investigator — Minneapolis Heart Institute
Locations (1):
- Minneapolis Heart Institute Foundation, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No